CLINICAL TRIAL: NCT06035159
Title: The Feasibility, Usability and Satisfaction of an Online Tool for the Treatment of Anxiety and Depressive Symptoms in the Perinatal Period (from Pregnancy to 1 Year After Delivery)
Brief Title: The Feasibility, Usability and Satisfaction of an Online Tool for Perinatal Mental Health Problems
Acronym: e-PMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: OnlinePsyHulp, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ONZ-2022-0386
Record Dates: First submitted 2023-07-26; First posted 2023-09-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depression; Depressive Disorder, Major; Depression, Postpartum; Anxiety; Anxiety Disorders; Pregnancy Related
Keywords: software, psychotherapy, telemedicine
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- online psychotherapy (Other): All participants have access to the psychotherapeutic intervention, which consists of 6 modules. Initially, we want to get information about the feasibility, comprehensibility and satisfaction of the participants with the tool. Secondly, the effectiveness of the intervention will be assessed through a pre-post measurement.
  Interventions: Behavioral: online psychotherapy

INTERVENTIONS:
Behavioral: online psychotherapy — 6 modules

SUMMARY:
With this study the investigators aim to examine through a mixed method study the feasibility, usability and satisfaction with the developed online tool for perinatal mental health problems. This will be done through a pre- and post measurement of depressive and anxiety symptoms and the use of the tool itself. In addition, a qualitative thematic analysis will be conducted on the clarity, understandability and user-friendliness of the tool.

DETAILED DESCRIPTION:
With the development and implementation of an online treatment tool, the existing online offer in Flanders (depression help, suicide) can be extended to pregnant women and women giving birth. This was necessary in the absence of a specific treatment offer for perinatal mental health problems.

In the framework of Project 2.0 of the Flemish Government, an online tool for the treatment of depressive and anxiety symptoms in the perinatal period has been developed by the Center for PMG UZ Gent (Mrs. Rita Van Damme, Prof. Dr. Gilbert Lemmens) in collaboration with the research group of Prof. Dr. Patrick Luyten (KUL). Online interventions have a wide reach, are easily accessible, have a destigmatizing effect and have a preventive function by reducing anxiety and depressive symptoms.

The online tool consists of 6 modules (parenting, relationships, self-care, emotions, cognitions and holding plan). It is recommended to do 1 module per week. The online tool will be launched in cooperation with OnlinePsyHulp, a GGZ group responsible for the website www.depressiehulp.be.

Through a mixed method study, the investigators aim to examine the feasibility, usability and satisfaction of the tool with a pre- and post measurement in preparation for a clinical trial. By means of an online application procedure, we will check whether participants applying to be enrolled in the study meet the inclusion criteria (pregnant woman or woman giving birth, partner of pregnant woman or woman giving birth, depressive or anxiety symptoms, 18 years or older, perinatal period (pregnancy to 1 year after birth), Dutch-speaking, living in Belgium). Participants meeting the inclusion criteria can enroll in the study after providing online informed consent, including email address.

At the start of the online tool, a number of demographic data (age, sex, marital status, education level, ethnicity, number of pregnancies, number of other (living) children, (expected) delivery date, current treatment modalities (medications, psychotherapeutic interventions, other), use of emotional support, psychiatric history) and questionnaires regarding depressive, anxiety and stress symptoms will be completed. These questionnaires, the Depression Anxiety Stress Scale (DASS 21-R) and the Edinburgh Postnatal Depression Scale (EPDS) will be repeated at follow-up (8 weeks after start). The question about other forms of treatment and use of emotional support will also be repeated at follow-up. The participant may receive up to 2 reminder emails (one per week) asking them to still complete these questionnaires after the online therapy. This should allow the researchers to calculate an effect through a pre-post measurement. In addition the investigators would like to conduct a qualitative thematic analysis on the feasibility, usability and satisfaction with the treatment program. This by means of the System Usability Scale (SUS) and 1 qualitative open-ended question on the usability of the tool (2 weeks after last login) and patient satisfaction after each lesson/module and 2 weeks after last login by means of qualitative questions (Likert scale and (open-ended) in-depth questions. When a participant does not log in for 2 weeks, an email is sent asking if they still intend to log in and if not to complete the qualitative questions. After this, a maximum of 1 reminder email may be sent.

Outcome measures are: 1) the reduction of depressive, anxiety and stress symptoms using DASS 21-R and EPDS (the latter to compare with other studies regarding depressive symptoms) after using the tool 2) the use of the online tool (via time logged in, number of logins and number of modules started, number of exercises completed), 3) the feasibility and understandability by the SUS and 1 qualitative open question regarding the usability of the tool 4) the determination of patient satisfaction through qualitative questions (Likert scale and (open-ended) in-depth questions.

ELIGIBILITY:
Inclusion Criteria:

* pregnant or giving birth
* partner of pregnant/birthing woman
* depressive or anxiety symptoms,
* 18 years or older,
* perinatal period (pregnancy up to 1 year after birth),
* Dutch-speaking,
* living in Belgium

Exclusion Criteria:

* younger than 18 years of age,
* outside perinatal period,
* do not speak Dutch well enough,
* not resident in Belgium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
use of the online tool, by means of time logged in | up to 10 weeks
  time spent logged in (minutes)
use of the online tool, by means of number of log-ins | up to 10 weeks
  number of log-ins (number)
use of the online tool, by means of number of lesson/modules started | up to 10 weeks
  number of modules started (number)
use of the online tool, by means of number of exercises completed | up to 10 weeks
  number of exercises completed (number)
usability of the online tool, by means of the System Usability Scale (SUS), when participant completes the program | through study completion, after each module (up to 10 wks)
  the system usability scale, the SUS, total score
usability of the online tool, by means of the System Usability Scale (SUS) when participant no longer logs in and after invitation through email reminder | 2 weeks
  the system usability scale, the SUS, total socre
usability of the online tool, by means of an open-ended qualitative question when participant completes the program. | through study completion, after each module (up to 10 wks)
  a qualitative open question
usability of the online tool, by means of an open-ended qualitative question, when participant no longer logs in and after invitation through email reminder | 2 weeks
  a qualitative open question
patient satisfaction, by means of qualitative questions when participant completes the program | through study completion, after each module (up to 10 wks)
  qualitative questions (Likert scale)
patient satisfaction, by means of open-ended qualitative questions, when participant completes the program | through study completion, after each module (up to 10 wks)
  qualitative questions (open-ended) in-depth questions
patient satisfaction, by means of qualitative questions when participant no longer logs in, and after invitation through email reminder | 2 weeks
  qualitative questions (Likert scale)
patient satisfaction, by means of open-ended qualitative questions when participant no longer logs in and after invitation through email reminder | 2 weeks
  qualitative questions (open-ended) in-depth questions.

SECONDARY OUTCOMES:
reduction of depressive, anxiety and stress symptoms as pre-measurement | baseline
  DASS 21-R, total score and scores of depressive scale (normal [0-9], mild [10-13], moderate [14-20], severe [21-27], extremely severe [28+]); anxiety scale (normal [0-7], mild [8-9], moderate [10-14], severe [15-19], extremely severe [20+]); stress scale (normal [0-14], mild [15-18], moderate [19-25], severe [26-33], extremely severe [34+]); Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.Scores on the DASS-21 will need to be multiplied by 2 to calculate the final score. The DASS-21 is based on a dimensional rather than a categorical conception of psychological disorder.
reduction of depressive, anxiety and stress symptoms as post-measurement | study completion (up to 10 weeks)
  DASS 21-R, total score and scores of depressive scale (normal [0-9], mild [10-13], moderate [14-20], severe [21-27], extremely severe [28+]); anxiety scale (normal [0-7], mild [8-9], moderate [10-14], severe [15-19], extremely severe [20+]); stress scale (normal [0-14], mild [15-18], moderate [19-25], severe [26-33], extremely severe [34+]); Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.Scores on the DASS-21 will need to be multiplied by 2 to calculate the final score. The DASS-21 is based on a dimensional rather than a categorical conception of psychological disorder.
reduction of depressive and anxiety symptoms as pre-measurement | baseline
  EPDS, total score (continuous and cut-off >= 13); EDS-3A(3 anxiety questions) (continuous and cut-off >= 5)
reduction of depressive, and anxiety symptoms as post-measurement | study completion (up to 10 weeks)
  EPDS total score (continuous and cut-off >= 13); EDS-3A (3 anxiety questions)(continuous and cut-off >= 5)

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Lemmens, Prof, Principal Investigator — University Hospital of Gent - University of Gent
Locations (1):
- University Hospital of Gent, Ghent, Belgium

REFERENCES:
- See also: online psychotherapy tool — http://depressiehulp.be/zelfhulp/zwangerschap